CLINICAL TRIAL: NCT04413474
Title: Does Ultrasonographic Assessment of Gastric Antrum Correlate With Gastric Residual Volume in Critically Ill Patients? A Prospective Study
Brief Title: Ultrasonographic Assessment of Gastric Residual Volume
Status: Completed | Type: Observational
Sponsor: Gurhan Taskin (Other)
Responsible Party: Sponsor-Investigator, Gurhan Taskin, Principal Investigator, Gulhane School of Medicine
Organization: Gulhane School of Medicine (Other)
Other Study IDs: 2017/72
Record Dates: First submitted 2020-05-23; First posted 2020-06-04 (Actual); Last update posted 2020-06-17 (Actual); Status verified 2020-06

CONDITIONS: Critically Ill; Enteral Feeding Intolerance
Keywords: critical care; ultrasonography; enteral feeding; enteral nutrition; feeding intolerance; gastric volume
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study group: Unselected critically ill patients who met the inclusion criteria

SUMMARY:
A recent systematic review reported that the prevalence of enteral nutrition intolerance in critically ill patients ranged from 2% to 75%, and the pooled rate was 38.3%.Many randomized controlled trials have reported that the incidence of pneumonia, regurgitation and aspiration do not correlate well with gastric residual volume (GRV) monitoring. In addition, it was reported that GRV monitoring may cause more frequent obstructions in the enteral tube access, leading to greater loss of time for intensive care unit nurses and patients receiving less than the prescribed daily intake due to enteral nutrition interruptions. The most recent SCCM/ASPEN guidelines in 2016 recommended that GRV monitoring not be included in the daily care protocol, but many institutions still use it to determine whether to continue enteral nutrition or to detect enteral tube-feeding intolerance. This study aimed to evaluate the relationship between ultrasonographic gastric antral measurements and aspirated gastric residual volume GRV in mechanically ventilated critically ill patients receiving enteral tube feeding via nasogastric, orogastric, or percutaneous gastrostomy tubes.

DETAILED DESCRIPTION:
Data collection and measurements:

The following clinical parameters of included patients will be recorded: age, sex, body weight, height, body mass index, Acute Physiology and Chronic Health Evaluation II (APACHE II) score on the day of admission,the Charlson Comorbidity Index score, any comorbid diseases, the total amount of EN product during the last 24 hours before ultrasonographic assessment, vasopressor therapy during imaging, and the dose of the vasopressors.

Ultrasonographic gastric antrum imaging procedure:

Ultrasonographic gastric antrum imaging will be carried out by the same intensivist on each patient just before routine tube-feed aspiration. Gastric antrum images will be obtained with a 2.5-6 MHz curvilinear probe placed in the sagittal plane of the epigastric region. All imaging attempts will be carried out in a 30-degree head-elevation supine position as described previously. Reference points will be used to obtain images of the gastric antrum-left anterior lobe of the liver, head of pancreas and abdominal aorta.The anteroposterior and craniocaudal diameters of the gastric antrum will be measured three times for each ultrasonographic assessment. The mean value of the three will be recorded. The universally accepted Two-Diameter Method defined by Bolondi et al. will be used for the measurement of antral cross-sectional area.

Tube-feeding aspiration (GRV measurement) procedure:

Routine gastric residual volume aspirations will be performed by the nursing staff blinded to the ultrasonographic measurements. The time between gastric antrum imaging and the beginning of GRV aspiration will be recorded in minutes. Gastric contents will slowly aspirated with 50 ml syringes for at least 10 minutes until stomach contents could no longer be aspirated. Patients will be reassessed with ultrasonography after the aspiration to ensure that the stomach is completely emptied with aspiration.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Mechanically ventilated in the intensive care unit
* Receiving enteral tube feeding via nasogastric, orogastric, or percutaneous gastrostomy tubes, and the tip of the enteral feeding-tube having been shown to be present in the stomach in a recent x-ray

Exclusion Criteria:

* Pregnancy
* Intestinal obstruction, gastric perforation, known upper gastrointestinal anatomical problem (e.g., hiatal hernia, gastric cancer, etc.)
* Food and liquid by mouth being withheld due to long-term fasting requirement for any medical reasons (e.g., gastrointestinal tract bleeding, etc.)

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mechanically ventilated critically ill patients receiving enteral feeding via nasogastric, orogastric, or percutaneous gastrostomy tubes who admitted to ICU in a one year period
Sampling Method: Probability Sample
Enrollment: 56 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2019-01-19 (Actual); Study Completion 2019-01-19 (Actual)

PRIMARY OUTCOMES:
Correlation between antral cross-sectional area and enteral tube feeding volumes. | From date of inclusion until the date of enteral tube-feeding termination or until the date of weaning from mechanical ventilation or until the date of discharging from ICU or until the date of the death, whichever came first, assessed up to one month.
  The correlation between aspirated tube-feeding volumes and ultrasonographic gastric antral cross-sectional area measurements in critically ill patients receiving enteral tube feeding.

CONTACTS AND LOCATIONS:
Overall Officials: Gurhan Taskin, MD, Principal Investigator — Gulhane School of Medicine
Locations (1):
- University of Health Sciences, Trabzon Kanuni Training and Research Hospital, Trabzon, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
All individual patient data that underlie results in a publication
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Starting 6 months after publication
Access Criteria: If requested the individual patient data will be shared.